CLINICAL TRIAL: NCT03613961
Title: Differential Effects of Propofol Induction Anaesthesia on the Heart Rate Variability Dynamics
Brief Title: Effects of Propofol Induction Anaesthesia on the Heart Rate Variability
Status: Completed | Type: Observational
Sponsor: National Central University (Other)
Responsible Party: Principal Investigator, Hsin-Yi Wang, Taipei Veterans General hospital, attending doctor of anesthesiology, National Central University
Other Study IDs: VGHTPE
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Autonomic Nervous System Imbalance
MeSH Terms: interventions — Anesthetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anesthetics — The ANS plays an important role in the regulation of hemodynamics during anesthesia. Manually blous of propofol during induction anesthesia is reported to reduce both sympathetic and parasympathetic tone; however, it is not clear whether the changes in heart rate variability are associated with propofol concentration. We will observe the relationship of anesthetics and HRV dynamics.

SUMMARY:
The ANS plays an important role in the regulation of hemodynamics during anesthesia. Manually blous of propofol during induction anesthesia is reported to reduce both sympathetic and parasympathetic tone; however, it is not clear whether the changes in heart rate variability are associated with propofol concentration.

DETAILED DESCRIPTION:
Because the ANS, especially the sympathetic nervous system, plays a major role in regulating cardiovascular homeostasis, knowledge of how anesthetic agents modify sympathetic activity is important for understanding subsequent cardiovascular responses.

Spectral analysis of heart rate variability (HRV) is a promising new approach, widely used, noninvasive technique to assess the autonomic indexes of neural cardiac control and has been correlated to the integrity and balance of the sympathetic and parasympathetic activation status. The presence of low-frequency (LF) and high-frequency (HF) oscillatory rhythms in the variability of the R-R interval (RRI) is well established. To date, it is believed that LF is mediated by the parasympathetic and sympathetic systems, whereas HF is mediated primarily by the parasympathetic system. There has been a lot of methodological analysis developed to evaluate the ANS function during anesthesia. In this study, Continuous Wavelet Transform (CWT), believed as a reliable and robust method to access cardiorespiratory dynamics of the ANS due to its adaptability and adjustability between spectral and temporal scale using a window of variable width, was used as a method for analyzing dynamic cardiovascular signals during anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* The subjects were selected from patients scheduled for surgery under general anesthesia.

Exclusion Criteria:

* recent administration of sedative or opioid drugs, emergency surgery and impairment of renal, hepatic, cardiac or respiratory function.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients scheduled for surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
HRV dynamics | 2 minutes
  Evaluate the changes in heart rate variability at different propofol concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, R.o.c, Taiwan

IPD SHARING:
Plan to Share IPD: No
all collected IPD, that underlie results in a publication

REFERENCES:
- [Derived] Wang HY, Lo MT, Chen KH, Mandell S, Chang WK, Lin C, Ting CK. Strong Early Phase Parasympathetic Inhibition Followed by Sympathetic Withdrawal During Propofol Induction: Temporal Response Assessed by Wavelet-Based Spectral Analysis and Photoplethysmography. Front Physiol. 2021 Sep 13;12:705153. doi: 10.3389/fphys.2021.705153. eCollection 2021. PMID 34588990